Protocol Title: Extracoporeal shock wave therapy (ESWT) for the treatment of detrusor underactivity/ underactive bladder (DU/UAB) — a single center, randomized,

double-blind, placebo-controlled, prospective study

IRB No.: 201900500A0

NCT No.: NCT04161183

Date: 2021-Jan-26

#### 7. STATISTICAL ANALYSIS

# 7.1. Evaluability

Patients receiving baseline screening and treatment will be considered as intent-to-treat (ITT) population. The ITT population with the following conditions will be considered as per-protocol (PP) population:

- 1. Not taking any prohibited medications
- 2. Fulfilling all entry criteria
- 3. Have treatment visit and post-treatment evaluations on the primary endpoint

The efficacy evaluation will be performed on both the ITT and PP datasets while the safety evaluations will be performed only on the ITT datasets. The primary conclusions will be made for the primary and secondary endpoints on the ITT patients.

## 7.2 Analysis

The statistical objective of this study is to demonstrate that the efficacy of ESWT is superior to placebo with respect to the decreases of UAB symptom score, and PVR. The safety profile of ESWT or placebo for the either group of treatment of patients with DU/UAB will also be confirmed.

## **Primary Efficacy Endpoint**

The efficacy of ESWT treatment will be evaluated for:

(1) Net changes of the mean post void residual (PVR) volume (mL) from baseline to 1 month after the treatment day.

## **Secondary Efficacy Endpoint**

The efficacy of ESWT will be evaluated for:

- (1) Net change of the following parameters from baseline to 1 month after the treatment day: functional bladder capacity (FBC), voiding frequency at daytime and voiding frequency at night time, incontinence, as record in 3-day voiding diary.
- (2) Global response assessment (GRA) of satisfaction by the patient (categorized into -3, -2, -1, 0, 1, 2, 3, indicating markedly worse to markedly improved) at 1 month after the treatment day. An improvement of GRA by 2 scales at 1 month is considered effective.
- (3) Net changes of the maximum flow rate, voided volume, Pdet@Qmax, and postvoid residual volume from baseline to 1 month after the treatment day.
- (4) Changes of Underactive Bladder Questionnaire (UAB-Q) score.
- (5) Changes of urinary nerve growth factor and cytokines level from baseline to 1 month after treatment day.

Voiding frequency at daytime and nighttime is measured as mean of the three-day voiding diary preceding the scheduled visit and the record days are 3 days.

Net change of each efficacy item will be analyzed by paired t-test between baseline and post-treatment in the treatment group and controlled group. The net changes of each efficacy item will be analyzed by ANOVA test to compare between treatment group and controlled groups. The global response assessment by the patients will be analyzed by Fisher exact test between the treatment and controlled groups.

All efficacy variables will be reported of respective point estimated and 95% confidence interval. Comparison tests will be reported of respective p value.

## **Secondary Safety Endpoints**

- (1) Local adverse event incidences (hematuria, micturition pain, UTI, urinary retention) will be reported by both treatment group and controlled group and by physiological systems as appropriate. Incidence of adverse events and the categories of adverse event severity between treatments will be analyzed. The coding system used will be COSTART.
- (2) The abnormalities of laboratory test results will be reported by patient list in the patients who have been tested for having severe adverse event.
- (3) The changes in physical examinations will be presented in the by-patient list.
- (4) All statistical tests used will be two-tailed with  $\alpha$ = 0.05.

# 7.3. Estimation of Incomplete Data

Due to this relatively small scale of clinical trial, any incomplete observation will be considered as missing data with no specific estimation for the incomplete data.

## 7.4 Sample Size

We used PASS 14 to calculate power for this study. Group sample sizes of 24 and 24 achieve 80.677% power to reject the null hypothesis of equal means when the population mean difference (Net changes of the mean post void residual (PVR) volume (mL) from baseline to 1 month after the treatment day) is -50.0 with a standard deviation for both groups of 60.0 and with a significance level (alpha) of 0.050 using a two-sided two-sample equal-variance t-test. According to 20% of the patient's drop-out rate, the number of subjects is set to 60, and the evaluator is 48 to get enough verification power.